CLINICAL TRIAL: NCT06401174
Title: Bridging the Gap: Delivering Equitable Colorectal Cancer Screening
Brief Title: Patient Navigation for Colorectal Cancer Screening
Acronym: SCREEN
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: National Committee for Quality Assurance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Screening
Other Study IDs: 6963
Record Dates: First submitted 2024-04-22; First posted 2024-05-06 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Cancer Screening
Keywords: disparities; Patient navigation

STUDY DESIGN:
Intervention Model Description: Step wedge trial with 5 six-month steps, three clinics at a time, for a total of 15 clinics.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient navigation (Experimental): Patient navigation will be rolled out at the clinic level (15 clinics). Referral orders will become available to participating clinics, with education and audit and feedback for providers. The study team will tailor patient navigation supports by clinic site for specifics on how the intervention is delivered.
  Interventions: Behavioral: Delivery of patient navigation
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Delivery of patient navigation — Clinics will receive educational materials and access a referral order for patient navigation. Iterative strategies will be used to increase CRC screening
  Arms: Patient navigation

SUMMARY:
Patient navigation is an evidence-based strategy to increase screening rates among racial and ethnic minorities, but there is a gap in understanding the multi-level influences on implementation of such programs across primary care practices. The investigators will conduct a stepped-wedge, randomized trial to roll out patient navigation and patient and provider reminders across 15 clinics (3 clinics per step, 5 six-month steps). Implementation strategies will include assessing for readiness, audit and feedback, building a community coalition, engaging consumers, modifying referral tracking, and training and educating clinical stakeholders. The research team will use the electronic health record data with consideration for the Observational Medical Outcomes Partnership (OMOP) Common Data Model, additional patient-reported data, and study tracking logs to measure reach, effectiveness, adoption, implementation, and will use qualitative measures and site observations to document contextual factors, including examination of discrimination in patient experiences and provider referral patterns that may influence intervention delivery or colorectal cancer screening completion.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) screening is recommended by the United States Preventative Services Task Force for adults age 45-75. Patient navigation is an evidence-based strategy to increase screening rates among racial and ethnic minorities. While patient navigation is an evidence-based approach to improve screening, there is a gap in understanding the multi-level influences on implementation of such programs across primary care practices, particularly using a health-equity focused, stakeholder-centered approach. Guided by the Practical, Robust Implementation and Sustainability Model (PRISM) and core health and racial equity principles, the investigative team aims to increase reach of patient navigation and show effectiveness through improvement in the percentage of Black and Hispanic patients completing CRC screening. Investigators will also utilize longitudinal tracking of implementation strategies to better track implementation or intervention adaptations navigation delivery in order to inform future scale up. The research team will conduct a stepped-wedged, randomized trial to roll out patient navigation and patient and provider reminders across 15 clinics (3 clinics per step, 5 six-month steps). Implementation strategies will include assessing for readiness, audit and feedback, building a community coalition, engaging consumers, modifying referral tracking, and training and educating clinical stakeholders. Researchers will use the electronic health record data with consideration for the Observational Medical Outcomes Partnership (OMOP) Common Data Model, additional patient-reported data, and study tracking logs to measure reach, effectiveness, adoption, implementation, and will use qualitative measures and site observations to document contextual factors, including examination of discrimination in patient experiences and provider referral patterns that may influence intervention delivery or CRC screening completion.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-75
* Due for colorectal cancer screening
* Identify as Black or Hispanic/Latino
* Attend primary care visit at one of the 15 selected clinics within the step time -period

Exclusion Criteria:

-

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Colorectal cancer screening completion | 12 months
  Completion of any USPSTF approved screening test

SECONDARY OUTCOMES:
Reach | 6 months
  Percent of patients referred out of those eligible
Adoption | 6 months
  Percent of providers referring to patient navigation
Acceptability measured by the Acceptability of Intervention Measure (AIM) | 12 months
  Stakeholder assessments of acceptability of navigation and implementation strategies measured on a four-item scale
Appropriateness measured by the Intervention Appropriateness Measure (IAM) | 12 months
  Stakeholder assessments of appropriateness of navigation and implementation strategies measured on a four-item scale
Feasibility measured by the Feasibility of Implementation Measure (FIM) | 12 months
  Stakeholder assessments of feasibility of navigation and implementation strategies measured on 4 item scale
Sustainability measured by the clinical sustainability assessment tool | 12 months
  Understanding clinical sustainability of interventions

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Internal Medicine Wisconsin Avenue, Washington D.C., District of Columbia
  - Family Medicine Spring Valley, Washington D.C., District of Columbia
  - Primary Care Lafayette, Washington D.C., District of Columbia
  - Family Medicine Fort Lincoln, Washington D.C., District of Columbia
  - Honeygo, Baltimore, Maryland
  - MedStar Adult Medicine at Union Memorial, Baltimore, Maryland
  - Harbor Hospital Primary Care Federal Hill, Baltimore, Maryland
  - Franklin Square, Baltimore, Maryland
  - Primary Care at Franklin Square, Baltimore, Maryland
  - Charlotte Hall, Charlotte Hall, Maryland
  - Internal Medicine Clinton, Clinton, Maryland
  - Family Medicine, Gaithersburg, Maryland
  - Internal Medicine Hyattsville, Hyattsville, Maryland
  - Family Medicine, Olney, Maryland
  - Olney Prof Park, Olney, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rivera Rivera JN, AuBuchon KE, Schubel LC, Starling C, Tran J, Locke M, Grady M, Mete M, Blumenthal HJ, Galarraga JE, Arem H. Supporting ColoREctal Equitable Navigation (SCREEN): a protocol for a stepped-wedge cluster randomized trial for patient navigation in primary care. Implement Sci Commun. 2024 Jun 3;5(1):60. doi: 10.1186/s43058-024-00598-5. PMID 38831365